CLINICAL TRIAL: NCT03758586
Title: An Efficient Single-Session Spatial Skill Trainer for Robot-assisted Surgery: A Randomized Trial
Brief Title: Spatial Skill Training for Robot-assisted Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0602-18-RMB
Record Dates: First submitted 2018-11-24; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Spatial Learning
MeSH Terms: conditions — Spatial Learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Surgical residents undergoing spatial skill training.
  Interventions: Other: Computerized spatial skill training
- Control group (Sham Comparator): Surgical residents not undergoing spatial skill training.
  Interventions: Other: Watching a presentation regarding robotic surgery

INTERVENTIONS:
Other: Computerized spatial skill training — The spatial skills training session consisted of six practice trials that were run in a sequence. The objective of each practice was to manipulate the simulated robotic arm to grab the cubes and move them to a desired location using keyboard keys. The participant was required to reach a decision based on the visual-spatial information, before initiating subsequent movements of the simulated robotic arm. Each practice trial presented an initial state of the cubes in front of the robotic arm, and a target position of the cubes.
  Arms: Study group
Other: Watching a presentation regarding robotic surgery — Watching a 20-35 minute long power-point presentation regarding the history of robotic surgery.
  Arms: Control group

SUMMARY:
Surgical residents from a single tertiary medical center were divided into 2 groups. All residents performed 2 tasks on a Da Vinci robotic simulator system after which they were either given a real training session in spatial skills (study group) or shown a short presentation regarding robotic surgery. After training/watching the presentation, they repeated the for mentioned tasks on the robotic simulator. Improvement in surgeon performance, especially regarding tissue damage was documented.

DETAILED DESCRIPTION:
Importance: Robot-assisted surgery is becoming the mainstay of modern surgery. Efficient training techniques are essential for enhanced performance. Optimal performance during a surgical task is key to successful surgery and minimal adverse events.

Objective: To introduce and examine a single session of spatial skill training as an efficient means of improving surgical suturing performance in robot-assisted surgery.

Design: Forty-one surgical residents will be randomly assigned to training and control conditions. (1) participants will perform two da-Vinci skills simulator (dVSS) tasks to determine baseline performance. (2) the training group will undergo computer-based simulator training of spatial skills while the control group will engage in a neutral activity. (3) two dVSS tasks will be performed within 2 days of training completion to evaluate post-training performance. The experiment will be conducted until December 2018.

Participants: A convenience sample comprised of 41 surgical residents with non-robotic surgical suturing skills.

ELIGIBILITY:
Inclusion Criteria:

* Surgical Residents with no previous robotic surgery experience.

Exclusion Criteria:

* Non surgical residents.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Tissue piercing | up to 2 hours from enrollment
  Number of times tissue was pierced during suturing
Tissue tearing | up to 2 hours from enrollment
  Number of times tissue was teared during suturing

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No